CLINICAL TRIAL: NCT02255305
Title: Fecal Microbiota Transplantation Versus Standard Medical Therapy for Initial Treatment of Recurrent Clostridium Difficile Infection
Brief Title: FMT Versus Antimicrobials for Initial Treatment of Recurrent CDI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to personnel issues for finding and enrolling patients, performing appropriate follow-up and performing FMT procedure
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Jennifer Grant, Hospital Epidemiologist, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH 14-331
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Clostridium Difficile Infection
Keywords: CDI; C difficile; C diff; Clostridium difficile
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Anti-Infective Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT Group (Intervention Arm) (Experimental): Patients randomized to the FMT group will have antimicrobials targeting C. difficile discontinued at least 6 hours prior to undergoing an FMT via retention enema. A second FMT via retention enema will be administered at 24 hours if diarrhea persists.
  Interventions: Biological: FMT
- Antimicrobial Group (Control Arm) (Active Comparator): Patients randomized to the antimicrobial group will be treated with antibiotics targeting C. difficile according to the Society for Healthcare Epidemiology of America (SHEA) Clinical Practice Guidelines for CDI. FMT will be offered to this group after 90 days if they experience relapsing CDI.
  Interventions: Drug: Antimicrobials

INTERVENTIONS:
Biological: FMT — Patients in the FMT group will receive ~50 grams of fecal material suspended in bacteriostatic normal saline and glycerol.
  Other Names: Fecal Microbiota Transplant; Stool Transplant
  Arms: FMT Group (Intervention Arm)
Drug: Antimicrobials — Patients randomized to the control group will receive antimicrobials targeting C. difficile.
  Arms: Antimicrobial Group (Control Arm)

SUMMARY:
The purpose of the study is to determine the safety and efficacy of Fecal Microbiota Transplant (FMT) for the treatment of the recurrence of Clostridium difficile infection (CDI) as compared to standard antibiotic therapy. Patients who have tested positive for CDI within 90 days of an admission for relapse of CDI will be approached to participate in this open-label, randomized controlled trial. Patients will either be randomized to the intervention group (receive FMT via retention enema) or the control group (receive antimicrobials targeting CDI).

DETAILED DESCRIPTION:
This trial is an open-label, randomized, controlled trial evaluating the safety and efficacy of fecal microbiota transplantation (FMT) for the treatment of the recurrence of Clostridium difficile infection (CDI) as compared to standard antibiotic therapy. Clostridium difficile infection (CDI) has increased in incidence and severity over the last decade and is associated with poor outcomes including increased morbidity, mortality, and healthcare costs (1-8). Relapse occurs in 15-35% of patients after the first episode of CDI and 45-65% of patients who have one relapse will experience a subsequent relapse (9, 10). Dysbiosis - decreased diversity of the fecal microbiome - is thought to contribute to the high rate of relapse (11). FMT quickly and successfully restores normal intestinal microorganisms of the diseased patient via infusion of a liquid stool preparation from a healthy donor. FMT resulted in disease resolution in ~90% of cases reported in a systematic review and meta-analyses without any significant adverse events noted (12, 13).

All hospitalized patients in the NorthShore system >18 years of age who are diagnosed with active CDI, defined as >3 diarrheal stools per day and a positive C. difficile polymerase chain reaction (PCR) assay, will be evaluated for inclusion in the study. Hospitalized patients presenting with their first or greater relapse of CDI occurring between 15 and 90 days after an index episode of CDI will be eligible for enrollment. Exclusion criteria will include pregnancy, neutropenia (absolute neutrophil count <1000/μl), contraindication for retention enema, or food allergy not controlled for in the donor diet. Eligible patients will undergo written informed consent followed by randomization into intervention and control groups.

Patients who are randomized to the intervention group will have antimicrobials targeting C. difficile discontinued at least 6 hours prior to undergoing an FMT via retention enema. A second FMT via retention enema will be administered at 24 hours if diarrhea persists. Patients randomized to the control group will be treated with antimicrobials targeting C. difficile according to the Society for Healthcare Epidemiology of America Clinical Practice Guidelines for CDI (18). FMT will be offered to the control group after 90 days if they experience relapsing CDI.

Two healthy "universal" donors who have previously donated fecal material for FMT have expressed willingness to participate in the study. Donors will complete the American Association of Blood Banks donor questionnaire for exposure to infectious agents as well as undergo serologic and stool testing for communicable diseases or pathogenic bacteria/viruses as previously described (17).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active C. difficile infection, defined as > 3 diarrheal stools per day and a positive C. difficile PCR assay
* Hospitalized patient presenting with first relapse of CDI occuring between 15 and 90 days after an index episode of CDI

Exclusion Criteria:

* Pregnancy
* Neutropenia (absolute neutrophil count <1000/microliters)
* Contraindication for retention enema
* Food allergy not controlled in the donor diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Becky Smith, MD, Principal Investigator — Endeavor Health; Jennifer Grant, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

REFERENCES:
- [Background] Dallal RM, Harbrecht BG, Boujoukas AJ, Sirio CA, Farkas LM, Lee KK, Simmons RL. Fulminant Clostridium difficile: an underappreciated and increasing cause of death and complications. Ann Surg. 2002 Mar;235(3):363-72. doi: 10.1097/00000658-200203000-00008. PMID 11882758
- [Background] Dubberke ER, Reske KA, Olsen MA, McDonald LC, Fraser VJ. Short- and long-term attributable costs of Clostridium difficile-associated disease in nonsurgical inpatients. Clin Infect Dis. 2008 Feb 15;46(4):497-504. doi: 10.1086/526530. PMID 18197759
- [Background] Kuijper EJ, Coignard B, Tull P; ESCMID Study Group for Clostridium difficile; EU Member States; European Centre for Disease Prevention and Control. Emergence of Clostridium difficile-associated disease in North America and Europe. Clin Microbiol Infect. 2006 Oct;12 Suppl 6:2-18. doi: 10.1111/j.1469-0691.2006.01580.x. PMID 16965399
- [Background] Loo VG, Poirier L, Miller MA, Oughton M, Libman MD, Michaud S, Bourgault AM, Nguyen T, Frenette C, Kelly M, Vibien A, Brassard P, Fenn S, Dewar K, Hudson TJ, Horn R, Rene P, Monczak Y, Dascal A. A predominantly clonal multi-institutional outbreak of Clostridium difficile-associated diarrhea with high morbidity and mortality. N Engl J Med. 2005 Dec 8;353(23):2442-9. doi: 10.1056/NEJMoa051639. Epub 2005 Dec 1. PMID 16322602
- [Background] McDonald LC, Owings M, Jernigan DB. Clostridium difficile infection in patients discharged from US short-stay hospitals, 1996-2003. Emerg Infect Dis. 2006 Mar;12(3):409-15. doi: 10.3201/eid1205.051064. PMID 16704777
- [Background] Musher DM, Aslam S, Logan N, Nallacheru S, Bhaila I, Borchert F, Hamill RJ. Relatively poor outcome after treatment of Clostridium difficile colitis with metronidazole. Clin Infect Dis. 2005 Jun 1;40(11):1586-90. doi: 10.1086/430311. Epub 2005 Apr 25. PMID 15889354
- [Background] Pepin J, Valiquette L, Alary ME, Villemure P, Pelletier A, Forget K, Pepin K, Chouinard D. Clostridium difficile-associated diarrhea in a region of Quebec from 1991 to 2003: a changing pattern of disease severity. CMAJ. 2004 Aug 31;171(5):466-72. doi: 10.1503/cmaj.1041104. PMID 15337727
- [Background] Brandt LJ, Aroniadis OC. An overview of fecal microbiota transplantation: techniques, indications, and outcomes. Gastrointest Endosc. 2013 Aug;78(2):240-9. doi: 10.1016/j.gie.2013.03.1329. Epub 2013 May 2. No abstract available. PMID 23642791
- [Background] Konijeti GG, Sauk J, Shrime MG, Gupta M, Ananthakrishnan AN. Cost-effectiveness of competing strategies for management of recurrent Clostridium difficile infection: a decision analysis. Clin Infect Dis. 2014 Jun;58(11):1507-14. doi: 10.1093/cid/ciu128. Epub 2014 Mar 31. PMID 24692533
- [Background] Chang JY, Antonopoulos DA, Kalra A, Tonelli A, Khalife WT, Schmidt TM, Young VB. Decreased diversity of the fecal Microbiome in recurrent Clostridium difficile-associated diarrhea. J Infect Dis. 2008 Feb 1;197(3):435-8. doi: 10.1086/525047. PMID 18199029
- [Background] Gough E, Shaikh H, Manges AR. Systematic review of intestinal microbiota transplantation (fecal bacteriotherapy) for recurrent Clostridium difficile infection. Clin Infect Dis. 2011 Nov;53(10):994-1002. doi: 10.1093/cid/cir632. PMID 22002980
- [Background] Kassam Z, Lee CH, Yuan Y, Hunt RH. Fecal microbiota transplantation for Clostridium difficile infection: systematic review and meta-analysis. Am J Gastroenterol. 2013 Apr;108(4):500-8. doi: 10.1038/ajg.2013.59. Epub 2013 Mar 19. PMID 23511459
- [Background] Hamilton MJ, Weingarden AR, Sadowsky MJ, Khoruts A. Standardized frozen preparation for transplantation of fecal microbiota for recurrent Clostridium difficile infection. Am J Gastroenterol. 2012 May;107(5):761-7. doi: 10.1038/ajg.2011.482. Epub 2012 Jan 31. PMID 22290405
- [Background] Youngster I, Sauk J, Pindar C, Wilson RG, Kaplan JL, Smith MB, Alm EJ, Gevers D, Russell GH, Hohmann EL. Fecal microbiota transplant for relapsing Clostridium difficile infection using a frozen inoculum from unrelated donors: a randomized, open-label, controlled pilot study. Clin Infect Dis. 2014 Jun;58(11):1515-22. doi: 10.1093/cid/ciu135. Epub 2014 Apr 23. PMID 24762631
- [Background] Kelly CR, Kunde SS, Khoruts A. Guidance on preparing an investigational new drug application for fecal microbiota transplantation studies. Clin Gastroenterol Hepatol. 2014 Feb;12(2):283-8. doi: 10.1016/j.cgh.2013.09.060. Epub 2013 Oct 6. PMID 24107393
- [Background] Cohen SH, Gerding DN, Johnson S, Kelly CP, Loo VG, McDonald LC, Pepin J, Wilcox MH; Society for Healthcare Epidemiology of America; Infectious Diseases Society of America. Clinical practice guidelines for Clostridium difficile infection in adults: 2010 update by the society for healthcare epidemiology of America (SHEA) and the infectious diseases society of America (IDSA). Infect Control Hosp Epidemiol. 2010 May;31(5):431-55. doi: 10.1086/651706. PMID 20307191

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm)
Started | 2 | 4
Completed | 1 | 0
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm) | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 89.5 (9.5) | 79.75 (24.9) | 83 (21.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Resolution of Diarrhea
Description: Number of patients with resolution of diarrhea and other abdominal symptoms or return to baseline symptoms that were present prior to C. difficile diagnosis
Time Frame: 90 days
Population: One patient in the control arm was lost to follow-up before the 30-day check in period
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm)
Number analyzed (Participants) | 2 | 3
Participants | 1 | 0

2. Secondary Outcome: Time to Clinical Resolution of Symptoms
Description: Amount of time it takes for patient to have cessation of diarrhea and abdominal pain/gastrointestinal symptoms (or return to baseline) and normalization of white blood cell count, creatinine, and temperature.
Time Frame: 90 days
Population: Unable to calculate time to clinical resolution as patients did not experience clinical resolution or lost to follow-up
Measure: Number; unit: days
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm)
Number analyzed (Participants) | 1 | 0
days | 44 |

3. Secondary Outcome: Hospital Length of Stay
Description: Patients' length of stay post-procedure will be measured
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm)
Number analyzed (Participants) | 2 | 4
days | 22 (18.4) | 6.5 (4.1)

4. Secondary Outcome: Number of Patients With Hospital Readmission
Description: Number of patients re-admitted to the hospital for recurrent Clostridium difficile infection
Time Frame: 90 days
Population: One patient in the control arm was lost to follow-up before the 30-day check in period
Measure: Number; unit: participants
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm)
Number analyzed (Participants) | 2 | 3
participants | 1 | 1

5. Secondary Outcome: Mortality
Description: Number of patients who died from any cause within 90 days of randomization
Time Frame: 90 days
Population: One patient in the control arm was lost to follow-up before the 30-day check in period
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm)
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | FMT Group (Intervention Arm) | Antimicrobial Group (Control Arm)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT Group (Intervention Arm) (N=2) | Antimicrobial Group (Control Arm) (N=4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (6) — Transient (< 24 hours) or intermittent nausea with no or minimal interference with oral intake
Fever (General disorders) | 0 (0) | 1 (1) — (99.9-100.5°F)
Diarrhea (Gastrointestinal disorders) | 2 (17) | 4 (17) — Transient or intermittent episodes of unformed stools OR Increase of ≤ 3 stools over baseline per 24-hour period
Fatigue/Malaise (General disorders) | 2 (18) | 4 (9) — Symptoms causing no or minimal interference with usual social & functional activities
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) — Transient or intermittent vomiting with no or minimal interference with oral intake
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Symptoms causing no or minimal interference with usual social & functional activities
Abdominal distention or bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (7)
Dehydration (General disorders) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0)
Colitis Symptoms (Gastrointestinal disorders) | 0 (0) | 0 (0)
Weight Loss (General disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Dysphagia (General disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study ended early due to personnel needed for study completion (enrollment, follow-up, FMT procedure) and did not reach enrollment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02255305/Prot_000.pdf